CLINICAL TRIAL: NCT03664713
Title: Efficacy of Eye Movement Desensitization and Reprocessing (EMDR) Therapy Compared to Treatment As Usual (TAU) in Psychiatric Inpatients With Severe Mental Disorder and a History of Psychological Trauma
Brief Title: EMDR in Psychiatric Inpatients With Severe Mental Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: EMDR Europe (Industry); Fundacion IMIM (Other)
Responsible Party: Principal Investigator, Ana Moreno Alcázar, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/7457/I
Record Dates: First submitted 2018-07-09; First posted 2018-09-10 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Severe Mental Disorder; Psychological Trauma
Keywords: Severe Mental Disorder; Psychological Trauma; Eye Movement Desensitization and Reprocessing Therapy
MeSH Terms: conditions — Mental Disorders; Psychological Trauma | interventions — Eye Movement Desensitization Reprocessing; Therapeutics

STUDY DESIGN:
Intervention Model Description: The project will be carried out in the sub-acute and long-stay inpatient wards of Parc de Salut Mar, Institute of Neuropsychiatry and Addiction (INAD), located in the Centre Forum. It consists of a single-blind RCT with two parallel branches, 1) individual therapy with EMDR and TAU, and 2) TAU only, with patients matched by age, sex, psychiatric diagnosis and premorbid IQ. Once the patient has been stabilized with psychotropic medication and has begun taking part in the psychosocial activities proposed by the unit, they will be offered the chance to receive 25 individual EMDR therapy sessions, each lasting 60 minutes. The patients will be evaluated at the beginning of their hospital stay, again when discharged from the unit and then at 6 and 12 month follow up.
Who Masked: Outcomes Assessor
Masking Description: Evaluators will be blind to treatment. Participants cannot be blind to treatment due to the impossibility of creating a sham alternative to EMDR therapy, due to its use of bilateral stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR plus TAU (Experimental): Individual Eye Movement Desensitization and Reprocessing (EMDR) Therapy: This consists of 25 individual sessions of 60 minutes each, applying the standard protocol with the existing validated modifications for specific pathologies. The standard EMDR protocol consists of 8 phases: 1) Patient history; 2) Patient preparation; 3) Evaluation of the main aspects of the traumatic memory; 4) Desensitization of the memory; 5) Installation of the positive cognition; 6) Body scan; 7) Close and 8) Reevaluation.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) Therapy
- TAU only (No Intervention): Treatment As Usual (TAU): The patients in this condition will participate in the psychosocial activities proposed by the inpatient unit (with a focus on autonomy, psychoeducation, treatment adherence, insight, functioning and family interventions). Patients who receive EMDR therapy will also participate in these activities.

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) Therapy — EMDR is an 8-phase psychological treatment composed of protocols and standardized procedures applicable to both adults and children. The eight phases (patient history, patient preparation, evaluation of the main aspects of the memory, desensitization of the traumatic memory, installation of the positive cognition, body scan, close and re-evaluation) and the protocol of the time line of past-present-future, allow a holistic evaluation of the image of the traumatic memory, and allow for the patient to be well-prepared before processing past events which underlie current pathology, current situations which cause perturbation, and challenges and possible future stimuli which might lead to the appearance of symptoms. (Shapiro, 2014)
  Arms: EMDR plus TAU

SUMMARY:
The study of psychological trauma has become increasingly important in the field of mental health research due to the strong negative impact it has on the course and prognosis of psychiatric pathologies. However, from a clinical point of view it is still an overlooked and even ignored component. There is scientific evidence that treating traumatic events at outpatient hospital services in patients with severe mental disorder improves both trauma-related symptoms and clinical symptoms. A first-line treatment for psychological trauma is Eye Movement Desensitization and Reprocessing (EMDR) therapy. This therapy is recommended by the World Health Organization for treating Post-Traumatic Stress Disorder and which has obtained promising first results in patients with severe mental disorder. This project proposes to test whether EMDR therapy in addition to standard treatment is more effective than standard treatment alone in psychiatric in-patients with severe mental disorder, in terms of reducing symptoms related to psychopathology and trauma, and in terms of improving functioning. Our first hypothesis is that EMDR will be more effective than standard treatment alone in reducing the severity of psychiatric symptoms. Our second hypothesis is that EMDR will be more effective than standard treatment alone in reducing the severity of trauma-related symptoms. Our third hypothesis is that EMDR will be more effective than standard treatment alone in improving functioning.

DETAILED DESCRIPTION:
Background

Severe mental disorders (SMD) are a group of diverse conditions which principally affect perception, cognition, emotion and behavioural control (Hyman et al. 2016). SMD has a significant health impact worldwide, both in economic terms as well as in mortality rate due to suicide or associated medical illnesses (Charlson et al. 2016), due to its high prevalence, frequent early age of onset, and its clinical course (usually chronic or with temporary improvements followed by relapse), and the cognitive deterioration of important mental capabilities.

The results of the different meta-analyses have shown that suffering adverse events in infancy significantly increases the risk of developing SMD in adult life (Bortolato et al., 2017; Palmier-Claus, Berry, Bucci, Mansell, & Varese, 2016). What is more, it is important to take into account that the presence of this comorbidity has important clinical implications, such as an increase in suicides, greater severity of symptoms, an increase in risky sexual behaviours, more hospital admissions, a worse disease course and a greater risk of being retraumatized (Rosenberg et al. 2007; Ford et al. 2007; Oquendo et al. 2005). However, at clinical level it is still an element which receives very little focus and may interfere in the correct evolution of the disease (Mauritz et al. 2013).

Two recently published studies in the severe psychiatric population have shown that the specific treatment of trauma improves in all cases the symptoms related to it in patients diagnoses with schizophrenia (van den Berg et al. 2015) and bipolar disorder (Novo et al. 2014), as well as showing an improvement in other clinical symptoms such as psychotic symptoms, paranoid ideation and hallucinations in the case of schizophrenia, and sub-syndromic symptoms in the case of bipolar disorder. In both studies, the intervention strategy used to treat traumatic events was EMDR (Eye Movement Desensitization and Reprocessing), a psychotherapeutic approach whose use in recent years has grown exponentially in clinical practice due to its great efficacy and safety, as well as being recommended by the World Health Organisation (WHO) and the American Psychiatric Association (APA) as a first line treatment for Post-traumatic Stress Disorder (PTSD) (Shapiro, 2014). It was developed at the beginning of the nineties by the North American psychologist Francine Shapiro to treat the consequences of psychological trauma. EMDR is an 8-phase psychological treatment composed of protocols and standardized procedures applicable to both adults and children. The eight phases (patient history, patient preparation, evaluation of the main aspects of the memory, desensitization of the traumatic memory, installation of the positive cognition, body scan, close and re-evaluation) and the protocol of the time line of past-present-future, allow a holistic evaluation of the image of the traumatic memory, and allow for the patient to be well-prepared before processing past events which underlie current pathology, current situations which cause perturbation, and challenges and possible future stimuli which might lead to the appearance of symptoms (Shapiro, 2014). The distinctive feature of this technique is the incorporation of bilateral stimulation, in the majority of cases through horizontal saccadic eye movements, into the combination of different theoretical and practical psychological orientations, in order to desensitize the suffering cause by traumatic memories and, as a consequence, achieve the reprocessing and the integration of these memories into the normalized biographic memories of the patient (Shapiro 2001). One of the main advantages of EMDR is that all protocols, both the standard and more specific ones, are standardized and scientifically validated both for clinical use and scientific scrutiny (Novo et al. 2016).

Evaluation & Diagnostic Protocol

In the baseline visit, sociodemographic data will be taken through a data collection notebook (CRD) and the validated Spanish versions of clinical, neuropsychological and trauma-related scales will be administered. Prior to discharge from the unit, the measures will be taken again, along with a measure regarding satisfaction of the treatment. Finally, all measures will be repeated at 6 and 12 months post-discharge as follow-up.

Side Effects and Follow Up

EMDR therapy is a safe and well tolerated psychological treatment. However, some may feel discomfort or suffer when the horizontal eye movements are carried out. If this occurs, bilateral stimulation will be achieved via tapping, which consists of small taps on the hands. Likewise, therapeutic work on difficult life experiences can accentuate psychological distress symptoms. The patient will be taught a variety of self-control techniques to be able to deal with the disturbing information which may arise during and between sessions. Any incident will be registered in the patient's clinical history as well as the CRD of the investigation project to later report the data.

Data Collection: Selection and Evaluation of Study Sample

Study participation is voluntary after being informed of the study objectives and having signed the informed consent document. The participants will be evaluated individually by specially trained health professionals (psychiatrists and psychologists qualified to make diagnoses). The project has been sent to the Ethical Committee for Clinical Investigations in Parc de Salut Mar for approval. Following the baseline evaluation, randomization will be carried out, stratified by age, sex and presence of prior trauma. Data will be collected after the EMDR sessions are finished, and participants will be contacted again at 6 months and 12 months follow up. Motives for refusal to participate in the study will be collected to determine the presence of selection bias in the sample and the causes of non-participation.

Statistical Analysis

Calculation of Sample Size: The study aims to evaluate the efficacy of the EMDR intervention protocol with TAU compared to TAU only in terms principally of clinical stabilization and improvement - a reduction in psychotic, anxiety, depressive and somatic symptoms amongst others. For this reason, the main variable will be the number of clinical relapses following the intervention, with a 12 month follow-up. Taking previous studies into account (Meyer & Hautzinger, 2012), the calculation of the size of the sample has been calculated based on a survival analysis with the statistical package "powerSurvEpi" for R (http://www.r-project.org) using an alpha of 0.005 instead of 0.05 to allow correction for multiple comparisons. The number of patients required to detect a hazard ratio = 2 in a Cox regression with a statistical power of 80% and an alpha of 0.005 is n=36 per intervention group (two groups: total n = 72). According to Chambless & Hollon (NO REFERENCE), a sample of this size should show clinically relevant differences. Assuming a dropout percentage of approximately 10-15% in trial patients, it will be necessary to recruit approximately 132 patients, 66 for each intervention condition.

Analysis of the main study variables The distribution of the between-group socio-demographic and clinical characteristics at baseline will be analysed using descriptive statistics. The continuous variables with a normal distribution will be analysed with a Multivariate Analysis of Variance (MANOVA). The change in clinical and biological variables compared to baseline at strategic times during the intervention will be analysed using an ANOVA with repeated measures including time factors, treatment conditions and their interaction. For cases which do not meet the normality premise, the Wilcoxon test will be used. The differences between groups, for the categorical and main clinical variables, will be analysed using the Chi-squared test. Those variables which are statistically significant can be used as covariables in a logistic or linear regression of the factors associated with the effect size, and to determine which variables are the best predictors of function. The effect size index will be estimated (Hedge's g or Pearson's r) for the correlation index of each analysis carried out. The statistical software used for all analyses will be the latest available version of SPSS (v. 24).

Analysis of Clinical Efficacy: For the main statistical analysis, the Intention to Treat (ITT) principal will be applied. The Last Observation Carried Forward (LOCF) will be used as the measure in cases of dropout.

Ethical Issues

The current Project will be carried out in accordance with the basic principles of protection of human rights and dignity as per the Helsinki Declaration and as per current legislation. The Law 14/2007 of Biomedical Investigation (LIB) will be followed for the biological samples. The study will not begin until the Ethical Committee for Clinical Investigations (CEIC) gives approval and all information gathered will be treated confidentially, as per constitutional law 15/1999, 13th December. Patients will be informed verbally and need to sign the attached informed consent.

Study limitations The fact that pharmacological treatment is not controlled for is a potential source of bias. To partially counteract this limitation, in the statistical analysis of the results the variable of pharmacological treatment will be taken into account.

Implications

The growing scientific interest in recent years regarding the impact of the presence of psychological trauma in the course and prognosis of mental disorders has demonstrated the great need to treat this risk factor from a clinical viewpoint, given the important negative consequences it means for patients. For this reason, and given the limited interest currently shown by the majority of mental health professionals, the investigators believe that proving the efficacy of implementing a trauma-focused treatment in an in-patient psychiatric setting is an innovative and pioneering proposal which can bring benefits not only to patients with psychotic symptoms, but also to the public health system through being cost-effective. This study has the potential to demonstrate the usefulness and the benefits of treating psychological trauma in psychiatric in-patients with clinical symptoms in a safe and effective way.

ELIGIBILITY:
Inclusion Criteria:

* sub-acute or long-stay ward in-patients diagnosed with an affective or non-affective psychotic disorder, as per DSM-V criteria, who also present a history of traumatic events.

Exclusion Criteria:

* abuse or dependence on substances in the previous 3 months (except nicotine), organic brain disease, presence of structured suicidal ideation and having received a trauma-focused therapy in the last 2 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Change in clinical severity from baseline to post-treatment at 6 months and follow up at 12 months. | The stated improvement will be seen at 6 months and maintained at 12 months.
  There will be a reduction in clinical severity of symptoms in the EMDR group as compared to the control group in terms of total score on the Brief Psychiatric Rating Scale (BPRS).

SECONDARY OUTCOMES:
Change in global clinical severity from baseline to post-treatment at 6 months and follow up at 12 months. | The stated improvement will be seen at 6 months and maintained at 12 months.
  There will be a reduction in global clinical severity in the EMDR group as compared to the control group as measured by the Clinical Global Impression Scale (CGI).
Change in depression symptoms from baseline to post-treatment at 6 months and follow up at 12 months. | The stated improvement will be seen at 6 months and maintained at 12 months.
  There will be a reduction in depression symptoms in the EMDR group as compared to the control group as measured by the Hamilton Depression Rating Scale (HDRS).
Change in mania symptoms from baseline to post-treatment at 6 months and follow up at 12 months. | The stated improvement will be seen at 6 months and maintained at 12 months.
  There will be a reduction in symptoms of mania in the EMDR group as compared to the control group as measured by the Young Mania Rating Scale (YMRS).
Change in symptoms of schizophrenia from baseline to post-treatment at 6 months and follow up at 12 months. | The stated improvement will be seen at 6 months and maintained at 12 months.
  There will be a reduction in symptoms related to schizophrenia in the EMDR group as compared to the control group as measured by the Positive and Negative Symptoms Scale (PANSS).
Change in number of patients with a Post-traumatic Stress Disorder (PTSD) diagnosis from baseline to post-treatment at 6 months and follow up at 12 months. | The stated improvement will be seen at 6 months and maintained at 12 months.
  Patients in the EMDR group will show a reduction in proportion of PTSD diagnosis as compared to the control group, as measured by the Global Evaluation of Posttraumatic Stress (EGEP-5).
Change in current impact of a traumatic event from baseline to post-treatment at 6 months and follow up at 12 months.. | The stated improvement will be seen at 6 months and maintained at 12 months.
  Patients in the EMDR group will show a reduced impact of a traumatic event as compared to the control group, as measured by the Impact of Events Scale-Revised (IES-R).
Change in number of dissociative symptoms from baseline to post-treatment at 6 months and follow up at 12 months. | The stated improvement will be seen at 6 months and maintained at 12 months.
  Patients in the EMDR group will show a reduced number of dissociative symptoms as compared to the control group, as measured by the Dissociative Experiences Scale (DES).
Change in global functioning from baseline to post-treatment at 6 months and follow up at 12 months. | The stated improvement will be seen at 6 months and maintained at 12 months.
  Patients in the EMDR group will show an improvement in their functional capacity as compared to the control group through the following scale: Functional Assessment Screening Tool (FAST), measuring the following areas: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Moreno-Alcázar, PhD, Principal Investigator — Parc de Salut Mar; Fundación IMIM; CIBERSAM.
Locations (1):
- Ana Moreno-Alcázar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Currently there are no plans.

REFERENCES:
- [Background] Shapiro F. The role of eye movement desensitization and reprocessing (EMDR) therapy in medicine: addressing the psychological and physical symptoms stemming from adverse life experiences. Perm J. 2014 Winter;18(1):71-7. doi: 10.7812/TPP/13-098. PMID 24626074
- [Background] Bortolato B, Kohler CA, Evangelou E, Leon-Caballero J, Solmi M, Stubbs B, Belbasis L, Pacchiarotti I, Kessing LV, Berk M, Vieta E, Carvalho AF. Systematic assessment of environmental risk factors for bipolar disorder: an umbrella review of systematic reviews and meta-analyses. Bipolar Disord. 2017 Mar;19(2):84-96. doi: 10.1111/bdi.12490. Epub 2017 May 3. PMID 28470927
- [Background] Ford JD, Hawke J, Alessi S, Ledgerwood D, Petry N. Psychological trauma and PTSD symptoms as predictors of substance dependence treatment outcomes. Behav Res Ther. 2007 Oct;45(10):2417-31. doi: 10.1016/j.brat.2007.04.001. Epub 2007 Apr 19. PMID 17531193
- [Background] Mauritz MW, Goossens PJ, Draijer N, van Achterberg T. Prevalence of interpersonal trauma exposure and trauma-related disorders in severe mental illness. Eur J Psychotraumatol. 2013;4. doi: 10.3402/ejpt.v4i0.19985. Epub 2013 Apr 8. PMID 23577228
- [Background] Novo Navarro P, Landin-Romero R, Guardiola-Wanden-Berghe R, Moreno-Alcazar A, Valiente-Gomez A, Lupo W, Garcia F, Fernandez I, Perez V, Amann BL. 25 years of Eye Movement Desensitization and Reprocessing (EMDR): The EMDR therapy protocol, hypotheses of its mechanism of action and a systematic review of its efficacy in the treatment of post-traumatic stress disorder. Rev Psiquiatr Salud Ment (Engl Ed). 2018 Apr-Jun;11(2):101-114. doi: 10.1016/j.rpsm.2015.12.002. Epub 2016 Feb 11. English, Spanish. PMID 26877093
- [Background] Novo P, Landin-Romero R, Radua J, Vicens V, Fernandez I, Garcia F, Pomarol-Clotet E, McKenna PJ, Shapiro F, Amann BL. Eye movement desensitization and reprocessing therapy in subsyndromal bipolar patients with a history of traumatic events: a randomized, controlled pilot-study. Psychiatry Res. 2014 Sep 30;219(1):122-8. doi: 10.1016/j.psychres.2014.05.012. Epub 2014 May 15. PMID 24880581
- [Background] Oquendo M, Brent DA, Birmaher B, Greenhill L, Kolko D, Stanley B, Zelazny J, Burke AK, Firinciogullari S, Ellis SP, Mann JJ. Posttraumatic stress disorder comorbid with major depression: factors mediating the association with suicidal behavior. Am J Psychiatry. 2005 Mar;162(3):560-6. doi: 10.1176/appi.ajp.162.3.560. PMID 15741474
- [Background] Palmier-Claus JE, Berry K, Bucci S, Mansell W, Varese F. Relationship between childhood adversity and bipolar affective disorder: systematic review and meta-analysis. Br J Psychiatry. 2016 Dec;209(6):454-459. doi: 10.1192/bjp.bp.115.179655. Epub 2016 Oct 6. PMID 27758835
- [Background] Rosenberg SD, Lu W, Mueser KT, Jankowski MK, Cournos F. Correlates of adverse childhood events among adults with schizophrenia spectrum disorders. Psychiatr Serv. 2007 Feb;58(2):245-53. doi: 10.1176/ps.2007.58.2.245. PMID 17287383
- [Background] van den Berg DP, de Bont PA, van der Vleugel BM, de Roos C, de Jongh A, Van Minnen A, van der Gaag M. Prolonged exposure vs eye movement desensitization and reprocessing vs waiting list for posttraumatic stress disorder in patients with a psychotic disorder: a randomized clinical trial. JAMA Psychiatry. 2015 Mar;72(3):259-67. doi: 10.1001/jamapsychiatry.2014.2637. PMID 25607833
- [Background] Charlson FJ, Baxter AJ, Dua T, Degenhardt L, Whiteford HA, Vos T. Excess Mortality from Mental, Neurological, and Substance Use Disorders in the Global Burden of Disease Study 2010. In: Patel V, Chisholm D, Dua T, Laxminarayan R, Medina-Mora ME, editors. Mental, Neurological, and Substance Use Disorders: Disease Control Priorities, Third Edition (Volume 4). Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2016 Mar 14. Chapter 3. Available from http://www.ncbi.nlm.nih.gov/books/NBK361935/ PMID 27227239
- [Background] Hyman S, Parikh R, Collins PY, Patel V. Adult Mental Disorders. In: Patel V, Chisholm D, Dua T, Laxminarayan R, Medina-Mora ME, editors. Mental, Neurological, and Substance Use Disorders: Disease Control Priorities, Third Edition (Volume 4). Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2016 Mar 14. Chapter 4. Available from http://www.ncbi.nlm.nih.gov/books/NBK361952/ PMID 27227248